CLINICAL TRIAL: NCT00271804
Title: Phase I Dose Escalation Trial of Bortezomib in Combination With Thalidomide in Patients With Myelodysplasia
Brief Title: Study of Velcade and Thalidomide in Patients With Myelodysplasia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: New study with lenalidomide pending
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Karen Ballen, Massachusetts general Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-381
Record Dates: First submitted 2005-12-30; First posted 2006-01-04 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic syndrome; Myelodysplasia; MDS; Velcade; Thalidomide; Bortezomib
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
The purpose of this study is to find out what the maximal tolerated dose of Velcade can be given with thalidomide in patients with myelodysplasia.

DETAILED DESCRIPTION:
Initial studies using Velcade in myelodysplasia with early results demonstrating that 35% had a partial response and 25% had stable disease. The combination of Velcade and thalidomide has been studied in patients with multiple myeloma, but not in patients with myelodysplasia. The CRR in the MM patients was 22%, with a good safety profile.

This is a phase 1, prospective, open-label, dose escalation study to evaluate the DLT and MTD of velcade with given in combination with thalidomide in patients with myelodysplasia. Treatment will be given as an outpatient. Patients will receive 4 days of Velcade (days 1, 4, 8, 11) and 21 days of thalidomide 50 mg/day for each 21 day cycle. There will be 3 cohorts of 3-6 patients each, plus 10 additional patients. The tree dose levels ill be 0.7, 1.0 and 1.3 mg/m2. Patients may continue to be treated up to 6 cycles. Cycles 2-6 will start within 2 weeks of completion of the previous cycle. Disease response will be evaluated after cycle 3 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Myelodysplastic syndrome with a IPSS score of 0.5 or greater
* May have had prior chemo/radiotherapy for another malignancy or myelodysplasia
* ECOG performance status of 0-2
* Life expectancy greater than 3 months
* Total bilirubin </+ 2xULN
* ALT and AST </+ 3xULN
* Calculated creatinine clearance > 30 ml/min
* Use of appropriate method of contraception during the study
* ANC > 0.5 x 10(9)
* Platelet count > 30 x 10(9)
* Consideration of treatment with 5 azacytidine is encouraged by not required

Exclusion Criteria:

* Ejection fraction < 40%
* myocardial infarction within 6 months of enrollment of New York Heart Association Class III or IV heart failure, uncontrolled angina, uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Women who are pregnant or breast-feeding
* Major surgery within 4 weeks prior to enrollment
* >/= grade 2 peripheral neuropathy within 14 days prior to enrollment
* Uncontrolled intercurrent illness
* Serious medical or psychiatric illness that could potentially interfere with the completion of treatment
* Hypersensitivity to bortezomib, boron, or mannitol
* Received an investigational drug within 14 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2005-06; Study Completion 2007-04

PRIMARY OUTCOMES:
The primary objective is to establish the maximally tolerated dose of bortezomib that can be administered with thalidomide in patient with myelodysplasia.

SECONDARY OUTCOMES:
Assess efficacy in terms of the number of patients attaining a 50% reduction in blast percentage, or 50% reduction in number of red blood cell and/or platelet transfusions.
Determine the toxicity profile of bortezomib when used in combination with thalidomide for patients with myelodysplasia.
Determine the relationship between NF-kB expression and clinical response to bortezomib and thalidomide.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ballen, M, Principal Investigator — Massachusetts General Hospital, Harvard University
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts